CLINICAL TRIAL: NCT00872469
Title: Tranexamic Acid for the Treatment of Postpartum Haemorrhage: An International Randomised, Double Blind, Placebo Controlled Trial
Brief Title: World Maternal Antifibrinolytic Trial
Acronym: WOMAN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ISRCTN76912190
Record Dates: First submitted 2009-03-30; First posted 2009-03-31 (Estimated); Last update posted 2018-02-26 (Actual); Status verified 2017-03

CONDITIONS: Postpartum Haemorrhage
Keywords: Postpartum haemorrhage; randomised controlled trial; tranexamic acid; antifibrinolytic
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Tranexamic Acid; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tranexamic acid (Active Comparator)
  Interventions: Drug: Tranexamic acid
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo [Saline]

INTERVENTIONS:
Drug: Tranexamic acid — 1-2 grams by intravenous injection
  Arms: Tranexamic acid
Drug: Placebo [Saline] — Matched to active comparator
  Arms: placebo

SUMMARY:
The WOMAN trial is a large pragmatic randomised double-blind, placebo controlled trial to quantify the effects of the early administration of tranexamic acid on death, hysterectomy and other relevant outcomes. 20,000 adult women, after delivery who have clinically diagnosed postpartum haemorrhage, are eligible if the responsible doctor is for any reason substantially uncertain whether or not to use an antifibrinolytic agent. Additionally, TWO nested studies will be conducted in a subset of women trial participants. The first nested study (ETAC) aims to evaluate the effect of tranexamic acid (TXA) on markers of coagulation in 400 women randomised to the WOMAN trial. The second nested study (ETAPLAT) aims to evaluate the haemostatic effect and antithrombotic effect of TXA in 128 women randomised to the WOMAN trial.

DETAILED DESCRIPTION:
BACKGROUND: Each year, worldwide about 530,000 women die from causes related to pregnancy and childbirth. Almost all (99%) of the deaths are in low and middle income countries. Obstetric haemorrhage is the leading cause of maternal mortality accounting for between one quarter and one third of deaths, most of which occur in the postpartum period. About 14 million mothers develop postpartum haemorrhage (PPH) each year and about 1-2% of them will die, with an average interval from onset to death of about 2 to 4 hours. Obstetric haemorrhage is also an important cause of maternal mortality in high income countries where it accounts for about 13% of maternal deaths.

Anti-fibrinolytic agents are widely used in surgery to reduce blood loss and the need for blood transfusion. A systematic review of randomised controlled trials of anti-fibrinolytic agents in elective surgery showed that tranexamic acid (TXA) reduced the risk of blood transfusion by a relative 39% (RR 0.61, 95% CI 0.54 to 0.69). In those requiring transfusion, TXA reduced the transfused blood volume by 1.1 units (95% CI 0.64 to 1.59). Anti-fibrinolytic agents also reduced the need for re-operation due to bleeding (RR=0.52: 95% CI 0.40 to 0.69). There was no evidence of an increased risk of thrombotic events.

TXA significantly reduces uterine blood loss in women with menorrhagia and is "recommended for consideration" as a treatment in intractable postpartum haemorrhage in the UK. However, at present there is little reliable evidence from randomised trials on the effectiveness of TXA in the treatment of PPH. A systematic review of randomised trials of TXA in PPH conducted by the applicants identified three trials of the prophylactic use of TXA, including a total of 460 participants. Although there was a significant reduction in average postpartum blood loss in women treated with TXA [weighted mean reduction 96 ml (95%CI 76ml to 109ml)] the quality of the trials was poor. None had adequate allocation concealment and even in aggregate the trials were too small to assess the effects of TXA on the clinically important end points of mortality, hysterectomy and thrombotic side effects. The most recently updated PPH treatment guidelines prepared by the World Health Organization (WHO) state that TXA may be used in the treatment of PPH if other measures fail, but points out that the quality of evidence on which this recommendation is based is low and recommends that further clinical trials of TXA in PPH are conducted.

AIM: The WOMAN Trial aims to determine the effect of the early administration of tranexamic acid (TXA) on death and hysterectomy in women with a clinical diagnosis of postpartum haemorrhage. The effect of TXA on the need for surgical interventions, blood transfusion, the risk of non-fatal vascular events (either haemorrhagic or occlusive), use of health services and breastfeeding will also be assessed.

OUTCOME: Outcomes will be collected at 42 days after randomisation, at discharge or at death (whichever occurs first).

TEST PRODUCT, DOSE AND MODE OF ADMINISTRATION: A first dose of Tranexamic acid (1 gram by intravenous injection) will be given as soon as possible after randomisation. If clinically indicated due to continued bleeding, a second dose of Tranexamic acid (1 gram by intravenous injection) will be given if within 4 hours of randomisation.

REFERENCE THERAPY, DOSE AND MODE OF ADMINISTRATION: A placebo (sodium chloride 0.9%) matched to the active drug will be administered in the same way as the active product. A placebo is justified in this trial because all women with PPH will receive all other treatments clinically indicated. Tranexamic acid/placebo will be given as an additional treatment.

SETTING: This trial will be co-ordinated from LSHTM and conducted in hospitals in low, middle and high income countries. It is likely that most patient recruitment will be in countries with high rates of mortality and morbidity from postpartum haemorrhage.

DURATION OF TREATMENT AND PARTICIPATION: The first dose will be given immediately after randomisation. If required, the second dose will be given up to 24 hours after randomisation. No further trial treatment will be given after 24 hours of randomisation. Participation will end at discharge, death or at 42 days post randomisation whichever occurs first.

CRITERIA FOR EVALUATION: All patients randomly assigned to one of the treatments will be analysed together, regardless of whether or not they completed or received that treatment on an intention to treat basis.

NESTED STUDY 1: Effect of tranexamic acid on coagulation in a sample of 400 participants in the WOMAN trial (ETAC). This aims to evaluate the effect of TXA on markers of coagulation in a sample of WOMAN trial participants. Standard coagulation parameters (platelets, ﬁbrinogen, PT and aPTT time and D-dimer) and ROTEM® parameters measured after in vitro activation with tissue factor (EXTEM) and inhibition with aprotinin (APTEM) will be determined (maximum lysis, maximum strength [Maximal Clot Firmness (MCF)], time from start to when the waveform reaches 2mm above baseline [Clotting Time (CT)], time from 2mm above baseline to 20mm above baseline [Clot Formation Time (CFT)], time to lysis [CLT (10% difference from MCF)], time to Maximum strength [MCF-t], Clot elasticity [MCE]).

NESTED STUDY 2: This aims to assess the haemostatic and antithrombotic effect of TXA in a sample of 128 participants in the WOMAN Trial (ETAPLAT). Platelet function, thrombin generation, fibrinogen level, D-Dimer and coagulation factors V, VIII and vWF will be assessed.

ELIGIBILITY:
All legally adult women with postpartum haemorrhage following vaginal or caesarean section delivery who have a clinical diagnosis of postpartum haemorrhage. The clinical diagnosis of PPH may be based on any of the following:

* Blood loss after vaginal delivery > 500 mL OR
* > 1,000 mL after caesarean section OR blood loss sufficient to compromise the haemodynamic status of the woman The fundamental eligibility criterion is the responsible clinician's 'uncertainty' as to whether or not to use an antifibrinolytic agent in a particular woman with postpartum haemorrhage.
* Women for whom the responsible doctor considers there is a clear indication for antifibrinolytic therapy should not be randomised.
* Women for whom there is considered to be a clear contraindication to antifibrinolytic therapy should not be randomised.

Where the responsible clinician is substantially uncertain as to whether or not to use an antifibrinolytic, all these women are eligible for randomisation and should be considered for the trial.

There are no other pre-specified exclusion criteria.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20060 (Actual)
Dates: Start 2009-05; Primary Completion 2016-06 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
The primary outcome is the proportion of women who die or undergo hysterectomy. The primary cause of death will be described. | up to 42 days after randomisation

SECONDARY OUTCOMES:
Surgical Interventions including hysterectomy; brace suture; selective arterial embolisation; laparotomy for other reasons; manual removal of placenta; intrauterine tamponade; artery ligation, to achieve haemostasis. | up to 42 days after randomisation
Need for blood transfusion - blood or blood component units transfused. | up to 42 days after randomisation
Health Status measured using the EQ-5D. | up to 42 days after randomisation
Thromboembolic events (myocardial infarction, strokes, pulmonary embolism, DVT). | up to 42 days after randomisation
Other relevant medical events | up to 42 days after randomisation
Length of stay at hospital/time spent at an intensive care unit | up to 42 days after randomisation
Need for mechanical ventilation. | up to 42 days after randomisation
Status of baby/ies | up to 42 weeks after randomisation of mother

OTHER OUTCOMES:
Primary outcome - ETAC - effect of TXA on fibrinolysis | 30 minutes after first dose is given
  Fibrinolysis will be measured with D-dimer, fibrinogen level and using ROTEM parameters previously reported to be associated with fibrinolysis (ie MCF, CA10, CA15, CLI30, and CLI60)
Secondary outcome - ETAC - Explore relationship between relationship between coagulation parameters and mortality | 42 days
Primary Outcome - ETAPLAT - effect of TXA on thrombin generation | 30 to 60 minutes after first dose is given
  (2) Thrombin Generation Assay [Lag Time (LT, min), peak height or time to peak (nMol) and area under the curve or endogenous thrombin potential (ETP, measured in nmol/L per min.)]
Secondary Outcome - ETAPLAT - TXA on platelet function, fibrinogen, D-Dimer and coagulation factor V, VIII and vWF levels | 30 to 60 minutes after first dose is given
  (1) Multiplate®tests (ADPtest and TRAPtest measured using AU per min) which will be performed with whole blood immediately after sampling. Fibrinogen level (Claus method, in g/L), D-Dimer (mg/L), Coagulation Factors V, VIII and vWF (measured with % of the norm) which will be performed on processed and separated platelet poor plasma

CONTACTS AND LOCATIONS:
Overall Officials: Ian G Roberts, MD, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- University College Hospital, Ibadan, Nigeria

IPD SHARING:
Plan to Share IPD: Yes
Will be available at https://ctu-app.lshtm.ac.uk/freebird/ in the future

REFERENCES:
- [Background] Shakur H, Elbourne D, Gulmezoglu M, Alfirevic Z, Ronsmans C, Allen E, Roberts I. The WOMAN Trial (World Maternal Antifibrinolytic Trial): tranexamic acid for the treatment of postpartum haemorrhage: an international randomised, double blind placebo controlled trial. Trials. 2010 Apr 16;11:40. doi: 10.1186/1745-6215-11-40. PMID 20398351
- [Derived] Kolin DA, Shakur-Still H, Bello A, Chaudhri R, Bates I, Roberts I. Risk factors for blood transfusion in traumatic and postpartum hemorrhage patients: Analysis of the CRASH-2 and WOMAN trials. PLoS One. 2020 Jun 3;15(6):e0233274. doi: 10.1371/journal.pone.0233274. eCollection 2020. PMID 32492040
- [Derived] Brenner A, Shakur-Still H, Chaudhri R, Fawole B, Arulkumaran S, Roberts I; WOMAN Trial Collaborators. The impact of early outcome events on the effect of tranexamic acid in post-partum haemorrhage: an exploratory subgroup analysis of the WOMAN trial. BMC Pregnancy Childbirth. 2018 Jun 7;18(1):215. doi: 10.1186/s12884-018-1855-5. PMID 29879947
- [Derived] Roberts I, Shakur H, Fawole B, Kuti M, Olayemi O, Bello A, Ogunbode O, Kotila T, Aimakhu CO, Olutogun T, Hunt BJ, Huque S. Haematological and fibrinolytic status of Nigerian women with post-partum haemorrhage. BMC Pregnancy Childbirth. 2018 May 9;18(1):143. doi: 10.1186/s12884-018-1794-1. PMID 29743045
- [Derived] WOMAN Trial Collaborators. Effect of early tranexamic acid administration on mortality, hysterectomy, and other morbidities in women with post-partum haemorrhage (WOMAN): an international, randomised, double-blind, placebo-controlled trial. Lancet. 2017 May 27;389(10084):2105-2116. doi: 10.1016/S0140-6736(17)30638-4. Epub 2017 Apr 26. PMID 28456509
- [Derived] Dallaku K, Shakur H, Edwards P, Beaumont D, Roberts I, Huque S, Delius M, Mansmann U. Statistical analysis plan for the WOMAN-ETAPlaT study: Effect of tranexamic acid on platelet function and thrombin generation. Wellcome Open Res. 2016 Dec 15;1:30. doi: 10.12688/wellcomeopenres.10105.2. PMID 28413832
- [Derived] Shakur H, Fawole B, Kuti M, Olayemi O, Bello A, Ogunbode O, Kotila T, Aimakhu CO, Huque S, Gregg M, Roberts I. Effect of tranexamic acid on coagulation and fibrinolysis in women with postpartum haemorrhage (WOMAN-ETAC): protocol and statistical analysis plan for a randomized controlled trial. Wellcome Open Res. 2016 Dec 16;1:31. doi: 10.12688/wellcomeopenres.10383.1. PMID 28317031
- [Derived] Shakur H, Roberts I, Edwards P, Elbourne D, Alfirevic Z, Ronsmans C. The effect of tranexamic acid on the risk of death and hysterectomy in women with post-partum haemorrhage: statistical analysis plan for the WOMAN trial. Trials. 2016 May 17;17(1):249. doi: 10.1186/s13063-016-1332-2. PMID 27188698
- See also: Trial website — http://www.womantrial.lshtm.ac.uk/
- See also: Sponsor — http://www.lshtm.ac.uk/